CLINICAL TRIAL: NCT02643953
Title: Increasing Women's Access to Skilled Pregnancy Care to Reduce Maternal and Perinatal Mortality in Nigeria: A Randomized Control Trial
Brief Title: Increasing Women's Access to Skilled Pregnancy Care to Reduce Maternal Mortality in Nigeria
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Sanni Yaya, Associate Professor, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 108041
Record Dates: First submitted 2015-12-28; First posted 2015-12-31 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Antenatal Care and Delivery
Keywords: Maternal Health; Maternal Mortality; Global Health; RCT
MeSH Terms: conditions — Maternal Death | interventions — Fertility; Residence Characteristics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (No Intervention): This arm includes women who are eligible and give birth (including cases of fetal or infant death) in the intervention period in comparative health wards, who will not receive the interventions and who will continue to receive their usual pattern of utilization of maternity care.
- Other (Experimental): The intervention will need to be multi-faceted, and will consist of provision of incentives to encourage women to attend primary health care and use family planning, antenatal, delivery and postnatal services; conditional cash transfers to promote uptake of services and targeted community health education and advocacy activities
  Interventions: Behavioral: Incentives; Behavioral: Community

INTERVENTIONS:
Behavioral: Incentives — 1) provision of incentives to encourage women to attend primary health care and use family planning, antenatal, delivery and postnatal services; 2) conditional cash transfers to promote uptake of services; 3) targeted community health education and advocacy activities; 4) community maternal audit/accountability activities, with community-led activities aimed at promoting utilization of services
  Arms: Other
Behavioral: Community — 1) outreach services by PHCs; 6) PHC strengthening including training of health providers; and 2) training and kitting of community health rangers who will be trained to follow up women at home to ensure that they do not default but that they continue to use PHC services until delivery.
  Arms: Other

SUMMARY:
Background: Nigeria has the second highest absolute number of maternal deaths and perinatal deaths in the world. The country contributes 14% of all maternal deaths worldwide, second only to India. Although all parts of the country are affected, most maternal, and perinatal deaths occur in the northeast and northwest geo-political zones, where women have limited access to evidence-based maternal and newborn health services. Affected women and families are mainly those who have little or no formal education, who are poor and marginalized, and who live in rural and sub-urban communities.

Problem: Research carried out in various regions of Nigeria has shown that insufficient access to pregnancy health services is a major factor that places women at high risk of adverse maternal and perinatal outcomes. Maternal care provided within Nigeria's numerous local Primary Health Centres (PHCs) is an efficient and practical avenue for reaching vulnerable women and their newborn infants, and PHC use is strongly encouraged by the Nigerian Federal Ministry of Health.

Research Question and Objective: The key research question and objectives are as follows: 1) To determine the main factors that prevent vulnerable women from using PHCs or receiving maternal and neonatal care therein; 2) To identify effective community level interventions for improving women's access to maternal health services, as a means to reduce maternal and perinatal morbidity and mortality in Nigeria.

Methodology: This study will complete a community-based, multi-site project using a mixed methods approach. The project will be done in three sequential phases: A data gathering phase (Phase 1), an intervention phase (Phase 2), and the implementation of the findings (Phase 3). The study will be conducted over 54-months in six communities, and another six communities of similar status will serve as control sites. During Phases 1-3, surveys about maternal health services utilization will be carried out at baseline, midterm and completion points of the project.

Potential Impact: Increasing women's access to evidence-based maternity care is likely a direct way to reduce maternal and neonatal mortality in Nigeria. The proposed project will determine how we can effectively increase access to PHCs, and then bring those findings into a policy and program format that can be applied across the country.

DETAILED DESCRIPTION:
Intervention Design: This intervention will be a randomized cluster trial design: interventions will be implemented in 6 health wards/communities (4 rural/peri-urban and 2 urban) while 6 health wards/communities with similar socio-demographic characteristics will serve as controls (where the intervention is not implemented). Including some urban or peri-urban clusters enables one to capture both rural and urban data about attitudes toward PMC maternal care (Phase 1), and the efficacy of the intervention to increase PMC use (Phase 2). It also enables one to see if attitudes (Phase 1 data) and the intervention (Phase 2) are different in rural vs. urban settings. This would be described as being a secondary analysis of the main data derived during Phase 1 and Phase 2.

The Intervention: The actual intervention activities to be applied will be finalized after the intervention workshop, following Phase 1. However, based on current knowledge, the intervention will need to be multi-faceted, and will possibly consist of 1) provision of incentives to encourage women to attend primary health care and use family planning, antenatal, delivery and postnatal services; 2) conditional cash transfers to promote uptake of services; 3) targeted community health education and advocacy activities; 4) community maternal audit/accountability activities, with community-led activities aimed at promoting utilization of services; 5) outreach services by PHCs; 6) PHC strengthening including training of health providers; and 7) training and kitting of community health rangers who will be trained to follow up women at home to ensure that they do not default but that they continue to use PHC services until delivery.

Control Group: The control group will comprise women who are eligible and give birth (including cases of fetal or infant death) in the intervention period in comparative health wards, who will not receive the interventions and who will continue to receive their usual pattern of utilization of maternity care. To ensure comparability of social, economic and cultural factors between the intervention and control groups, the health wards that will serve as controls will have been selected from the same States as the intervention health wards. Hence, the study will have paired intervention-control groups from the same States, but distanced enough from one another (in separate LGAs) to reduce the potential effects of study contamination (i.e., the intervention is known or adopted in a control region). However, should the intervention prove to be effective, the investigators will be recommending the use of the same intervention activities in the control sites, as well as throughout the country.

ELIGIBILITY:
Inclusion Criteria

1. Women who give birth (including cases of foetal or infant death) in comparative health wards and who receive their usual pattern of utilization of maternity care.
2. Women who have antenatal care record at one of the study facilities

Exclusion Criteria

1. Women outside the research regions who fail to meet any of the inclusion criteria will be excluded
2. Women who do not have an antenatal care record at one of the study facilities

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2020-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
The main outcome variable will be the proportion of women, among those who give birth following the start of the intervention, who use PHCs for antenatal, delivery and postnatal care, in the intervention and control health wards. | Up to 48 months

SECONDARY OUTCOMES:
A secondary outcome will be the proportion of women giving birth and attending PHCs who have received standard/quality antenatal, intrapartum and postnatal care. | Up to 48 months

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Harrison KA. The struggle to reduce high maternal mortality in Nigeria. Afr J Reprod Health. 2009 Sep;13(3):9-20. PMID 20690258
- [Background] Harrison KA. Are traditional birth attendants good for improving maternal and perinatal health? No. BMJ. 2011 Jun 14;342:d3308. doi: 10.1136/bmj.d3308. No abstract available. PMID 21673000
- [Background] Hogan MC, Foreman KJ, Naghavi M, Ahn SY, Wang M, Makela SM, Lopez AD, Lozano R, Murray CJ. Maternal mortality for 181 countries, 1980-2008: a systematic analysis of progress towards Millennium Development Goal 5. Lancet. 2010 May 8;375(9726):1609-23. doi: 10.1016/S0140-6736(10)60518-1. Epub 2010 Apr 9. PMID 20382417
- [Background] Lassi ZS, Bhutta ZA. Community-based intervention packages for reducing maternal and neonatal morbidity and mortality and improving neonatal outcomes. Cochrane Database Syst Rev. 2015 Mar 23;2015(3):CD007754. doi: 10.1002/14651858.CD007754.pub3. PMID 25803792
- [Background] Montoya A, Calvert C, Filippi V. Explaining differences in maternal mortality levels in sub-Saharan African hospitals: a systematic review and meta-analysis. Int Health. 2014 Mar;6(1):12-22. doi: 10.1093/inthealth/iht037. Epub 2014 Feb 18. PMID 24550236
- [Background] Moyer CA, Dako-Gyeke P, Adanu RM. Facility-based delivery and maternal and early neonatal mortality in sub-Saharan Africa: a regional review of the literature. Afr J Reprod Health. 2013 Sep;17(3):30-43. PMID 24069765
- [Background] Buor D, Bream K. An analysis of the determinants of maternal mortality in sub-Saharan Africa. J Womens Health (Larchmt). 2004 Oct;13(8):926-38. doi: 10.1089/jwh.2004.13.926. PMID 15671708
- [Background] Chinkhumba J, De Allegri M, Muula AS, Robberstad B. Maternal and perinatal mortality by place of delivery in sub-Saharan Africa: a meta-analysis of population-based cohort studies. BMC Public Health. 2014 Sep 28;14:1014. doi: 10.1186/1471-2458-14-1014. PMID 25263746
- [Background] Nkwo PO, Lawani LO, Ezugwu EC, Iyoke CA, Ubesie AC, Onoh RC. Correlates of poor perinatal outcomes in non-hospital births in the context of weak health system: the Nigerian experience. BMC Pregnancy Childbirth. 2014 Sep 30;14:341. doi: 10.1186/1471-2393-14-341. PMID 25271134
- [Background] Fapohunda B, Orobaton N. Factors influencing the selection of delivery with no one present in Northern Nigeria: implications for policy and programs. Int J Womens Health. 2014 Jan 31;6:171-83. doi: 10.2147/IJWH.S54628. eCollection 2014. PMID 24516341
- [Background] Aremu O, Lawoko S, Dalal K. Neighborhood socioeconomic disadvantage, individual wealth status and patterns of delivery care utilization in Nigeria: a multilevel discrete choice analysis. Int J Womens Health. 2011;3:167-74. doi: 10.2147/IJWH.S21783. Epub 2011 Jul 4. PMID 21792338
- [Background] Adamu YM, Salihu HM. Barriers to the use of antenatal and obstetric care services in rural Kano, Nigeria. J Obstet Gynaecol. 2002 Nov;22(6):600-3. doi: 10.1080/0144361021000020349. PMID 12554244
- [Background] Bhutta ZA, Ali S, Cousens S, Ali TM, Haider BA, Rizvi A, Okong P, Bhutta SZ, Black RE. Alma-Ata: Rebirth and Revision 6 Interventions to address maternal, newborn, and child survival: what difference can integrated primary health care strategies make? Lancet. 2008 Sep 13;372(9642):972-89. doi: 10.1016/S0140-6736(08)61407-5. PMID 18790320
- [Background] Rosato M, Laverack G, Grabman LH, Tripathy P, Nair N, Mwansambo C, Azad K, Morrison J, Bhutta Z, Perry H, Rifkin S, Costello A. Community participation: lessons for maternal, newborn, and child health. Lancet. 2008 Sep 13;372(9642):962-71. doi: 10.1016/S0140-6736(08)61406-3. PMID 18790319
- [Background] Lassi ZS, Haider BA, Bhutta ZA. Community-based intervention packages for reducing maternal and neonatal morbidity and mortality and improving neonatal outcomes. Cochrane Database Syst Rev. 2010 Nov 10;(11):CD007754. doi: 10.1002/14651858.CD007754.pub2. PMID 21069697
- [Background] Okonofua F, Lambo E, Okeibunor J, Agholor K. Advocacy for free maternal and child health care in Nigeria--Results and outcomes. Health Policy. 2011 Feb;99(2):131-8. doi: 10.1016/j.healthpol.2010.07.013. Epub 2010 Aug 19. PMID 20727612
- [Background] Lewycka S, Mwansambo C, Kazembe P, Phiri T, Mganga A, Rosato M, Chapota H, Malamba F, Vergnano S, Newell ML, Osrin D, Costello A. A cluster randomised controlled trial of the community effectiveness of two interventions in rural Malawi to improve health care and to reduce maternal, newborn and infant mortality. Trials. 2010 Sep 17;11:88. doi: 10.1186/1745-6215-11-88. PMID 20849613
- [Background] Thaddeus S, Maine D. Too far to walk: maternal mortality in context. Soc Sci Med. 1994 Apr;38(8):1091-110. doi: 10.1016/0277-9536(94)90226-7. PMID 8042057
- [Background] O'Donnell O. Access to health care in developing countries: breaking down demand side barriers. Cad Saude Publica. 2007 Dec;23(12):2820-34. doi: 10.1590/s0102-311x2007001200003. PMID 18157324
- [Background] Huda FA, Ahmed A, Ford ER, Johnston HB. Strengthening health systems capacity to monitor and evaluate programmes targeted at reducing abortion-related maternal mortality in Jessore district, Bangladesh. BMC Health Serv Res. 2015 Sep 28;15:426. doi: 10.1186/s12913-015-1115-6. PMID 26416690
- [Derived] Yaya S, Okonofua F, Ntoimo L, Kadio B, Deuboue R, Imongan W, Balami W. Increasing women's access to skilled pregnancy care to reduce maternal and perinatal mortality in rural Edo State, Nigeria: a randomized controlled trial. Glob Health Res Policy. 2018 Apr 4;3:12. doi: 10.1186/s41256-018-0066-y. eCollection 2018. PMID 29632896